CLINICAL TRIAL: NCT06757491
Title: Low-frequency Repetitive Transcranial Magnetic Stimulation Attenuates Visceral Pain in Irritable Bowel Syndrome With Diarrhea Via Inhibition of the Medial Prefrontal Cortex
Brief Title: Lf-rTMS Attenuates Visceral Pain in Irritable Bowel Syndrome With Diarrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-KY-08; BE2023710 (Other Grant/Funding Number: Jiangsu Provincial Department of Science and Technology)
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Repetitive Transcranial Magnetic Stimulation; Chronic Visceral Pain; Functional Magnetic Resonance Imaging; IBS (Irritable Bowel Syndrome); Clinical Efficacy
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham rTMS Group (Sham Comparator): For the sham rTMS group, the coil was placed over the mPFC with the rTMS function disabled, and pre-recorded acoustic artifacts were played to mimic the auditory experience of the rTMS group.
  Interventions: Device: Sham (No Treatment)
- rTMS Group (Active Comparator): Low-frequency rTMS (1 Hz) was applied to the mPFC using a TMS stimulator at 80% resting motion threshold intensity.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — A figure-of-eight coil is used to apply active low-frequency (1 Hz) rTMS to the corresponding representation area of theprefrontal cortex (mPFC). The treatment is administered for 20 minutes daily for a total of 2 weeks.
  Arms: rTMS Group
Device: Sham (No Treatment) — For the sham rTMS group, the coil was placed over the mPFC with the rTMS function disabled, and pre-recorded acoustic artifacts were played to mimic the auditory experience of the rTMS group.
  Arms: Sham rTMS Group

SUMMARY:
Objectives: To identify a central hub of visceral pain in IBS-D and elucidate the mechanism by which repetitive transcranial magnetic stimulation (rTMS) confers analgesic effects.

Methods: A total of 42 IBS-D patients were recruited and randomly assigned (1:1) to the sham rTMS or the rTMS group. A nested cohort of 21 IBS-D participants who completed baseline fMRI assessments prior to randomization was included. Consistent with the randomization procedure，these individuals were evenly distributed between the two groups. Both participants and outcome assessors remained blinded to treatment allocation throughout the study. All patients completed the two-week intervention and were included in the final analysis.

DETAILED DESCRIPTION:
Background：Chronic visceral pain in irritable bowel syndrome with diarrhea (IBS-D) is a profound therapeutic challenge. While aberrant central processing is implicated, the key brain regions driving this visceral pain and their suitability as neuromodulatory targets remain undefined.

Methods: Participants were randomly assigned (1:1) to the sham rTMS or rTMS group using a computer-generated randomization sequence created by an independent researcher who was not involved in recruitment, treatment, or outcome assessment. Allocation concealment was ensured using sequentially numbered, opaque, sealed envelopes, which were opened only after baseline evaluations were completed.

Both participants and outcome assessors were blinded to treatment allocation. The rTMS operators were not involved in data collection or analysis. For the sham condition, the coil was positioned identically over the mPFC with magnetic output disabled, and prerecorded clicking sounds were delivered to mimic the acoustic sensation of stimulation. Participants were asked not to discuss treatment sensations with assessors. Scale raters and fMRI analysts remained blinded until all analyses were finalized.

For the nested fMRI cohort, randomization and blinding procedures were identical, with group allocation revealed only after preprocessing and statistical analysis had been completed.

ELIGIBILITY:
All diagnoses were made by board-certified gastroenterologists. Eligible participants met the following inclusion criteria: (1) age between 18 and 75 years; (2) fulfillment of the Rome IV diagnostic criteria for IBS-D. Exclusion criteria included: (1) presence of inflammatory or other organic gastrointestinal diseases; (2) diagnosed psychiatric disorders; (3) history of anorectal, intestinal, or abdominal surgery; (4) pregnancy or lactation; (5) presence of metallic implants or cardiac pacemakers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Visceral Sensitivity Index | 2 weeks of treatment
  (1) Clinical control: After the course of treatment, clinical symptoms disappear; (2) Significant effect: After the course of treatment, the symptom grading is reduced by 2 levels; (3) Effective: After the course of treatment, the symptom grading is reduced by 1 level; (4) Ineffective: After treatment, those who do not meet the above standards.

SECONDARY OUTCOMES:
IBS-symptom severity score | 2 weeks of treatment
  The criteria were based on the IBS Symptom Severity Score (IBS-SSS), a hierarchical efficacy assessment method.The IBS-SSS consists of five entries assessing the degree of abdominal pain and discomfort, frequency of bdominal pain episodes, the degree of abdominal distension and discomfort, the degree of satisfaction with bowel habits and behaviors, and the degree of impact of intestinal symptoms on life,with a total score of 500 points. A score of 75-175 is considered mild, 176-300 is moderate, and over 300 is severe. Cure was defined as a total IBS symptom severity of less than 75; efficacy was defined as 2-level improvement in total score(e.g., symptoms improved from severe to mild); validity was defined as a 1-level improvement in tatal(e.g., symptoms improved from severe to moderate or symptoms from moderate to mild); and invalidity was defined as no improvement or deterioration in total score.

OTHER OUTCOMES:
anorectal manometry | 2 weeks of treatment
  Anorectal manometry was performed on the subjects before and after treatment and the subjects' rectal primary sensory thresholds were recorded. Rectal initial sensory thresholds between 20-90ml were considered normal , less than 20ml was considered as sensitivity rectal sensory, and cure meant that the IBS patients had their rectal initial sensory recordings restored to between 20-90ml.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Li, Dr., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
This clinical research protocol is just beginning to be studied at this time and sharing is not recommended at this time.